CLINICAL TRIAL: NCT00874692
Title: Randomised Controlled Trial of Boiler Management Systems in Social Housing in Camden: An Assessment of Health, Environmental and Economic Outcomes
Brief Title: Health and Environmental Effects of Boiler Management Systems in Social Housing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Camden Primary Care Trust, London (Unknown); London Borough of Camden Housing and Adult Social Care Directorate (Unknown)
Responsible Party: Dr. Phil Edwards, London School of Hygiene & Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: EPNPPT84
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-06

CONDITIONS: Hot Water Burns (Scalds)
Keywords: tap water temperature; social housing; scald reduction; Temperature (degrees Celsius) of hot tap water at point of delivery.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BMS and sterilisation (Experimental): BMS and sterilisation programme will be delivered
  Interventions: Other: BMS and sterilisation programme
- BMS standard water heating (No Intervention)

INTERVENTIONS:
Other: BMS and sterilisation programme — BMS with reduced hot water temperature and sterilisation programme
  Arms: BMS and sterilisation

SUMMARY:
The purpose of this study is to evaluate the impact of a passive safety measure, namely a reduction in centrally controlled hot tap water temperatures in social housing using a boiler management system, as an effective public health intervention.

DETAILED DESCRIPTION:
The annual hospital admission rate in England for burns and scalds is 31 children per 100,000 population. While reducing the temperature in domestic hot water tanks is a recommended injury prevention strategy, the UK has been slow to adopt such 'passive' safety measures. However, Camden Council employs a Boiler Management System (BMS) in boiler houses to centrally set the hot water temperature for parts of its social housing stock, providing the opportunity to evaluate various impacts of a 'passive' safety measure, including quantifying the effects of the BMS on average hot water temperatures at delivery, annual energy costs, and annual greenhouse gas emissions; modelling the reduction in scald injuries; identifying the cost-effectiveness of the system as a public health intervention; as well as describing experiences/ perceptions of risk of scalding and identifying health and social benefits of the BMS. Boiler houses with BMS will be randomised to remain at their constant set temperature or to BMS reduced temperature and sterilisation programme. A process evaluation will also be undertaken to assess the acceptability of water temperatures to tenants.

ELIGIBILITY:
Inclusion Criteria:

* Individuals living in social housing in the London Borough of Camden where the Boiler Management system has been installed.

Exclusion Criteria:

* Aged under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Thermal energy (degrees Celsius) at hot tap of bath | after 1 minute

SECONDARY OUTCOMES:
Acceptability of hot water temperature delivered to tenant | Up to 2-3 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Phil Edwards, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Camden, London, United Kingdom

REFERENCES:
- [Derived] Edwards P, Durand MA, Hollister M, Green J, Lutchmun S, Kessel A, Roberts I. Scald risk in social housing can be reduced through thermostatic control system without increasing Legionella risk: a cluster randomised trial. Arch Dis Child. 2011 Dec;96(12):1097-102. doi: 10.1136/archdischild-2011-300606. Epub 2011 Sep 20. PMID 21937486